CLINICAL TRIAL: NCT00327743
Title: A Dose-escalating, Multicenter, Single Arm, Open-Label Study of XRP9881 in Combination With Capecitabine (Xeloda), in Metastatic Breast Cancer Patients With Disease Progressing After Anthracycline and Taxane Therapy
Brief Title: Combination Study of a New Taxane and Capecitabine in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD6511; EudraCT:2006-006474-21
Record Dates: First submitted 2006-05-04; First posted 2006-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer; Cancer
Keywords: Cancer Alternative Therapies; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — larotaxel; Capecitabine

ARMS (1):
- larotaxel + Capecitabine (Experimental)
  Interventions: Drug: larotaxel; Drug: capecitabine

INTERVENTIONS:
Drug: larotaxel — IV infusion on Day 1 of a 21-day cycle
  Other Names: XRP9881
Drug: capecitabine — oral, twice daily, Day 1-Day 14 of a 21-day cycle

SUMMARY:
The goal of this phase I-II clinical research study is to find the highest safe dose of XRP9881 and capecitabine that can be given in combination in the treatment of metastatic breast cancer in patients who have been previously treated by taxanes and anthracyclines. The safety and effectiveness of this combination will also be studied. Patients participating in the study will be asked to give additional blood samples to look at the level of study drugs in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast adenocarcinoma that is now metastatic or locally recurrent and inoperable with curative intent.
* Prior treatment with a standard regimen of anthracycline and taxane.
* Female patients at least 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-2
* Adequate organ and bone marrow function
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (For the part I component, patients with non-measurable disease are accepted.)
* Resolution of all clinically significant toxic effects
* Completion of all prior therapy ≥ 3 weeks prior to registration. Patients on bisphosphonate therapy may continue such therapy.
* Patients must be either post-menopausal, surgically sterile, or using effective contraception.
* Willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

* History of any second malignancy within the last 5 years (except adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri).
* Patients receiving more than one adjuvant regimen or more than one metastatic regimen
* Known brain or leptomeningeal disease.
* Concurrent treatment on another clinical trial or with any other cancer therapy including chemotherapy, biological therapy, hormonal therapy, radiotherapy, chemoembolization therapy, cryotherapy, targeted non-cytotoxic therapies, or patients planning to receive these treatments during the study.
* Prior treatment with capecitabine, XRP9881, or any investigational chemotherapy.
* History of hypersensitivity to taxanes, Polysorbate-80, or to compounds with similar chemical structures. Patients with known intolerance to fluoropyrimidines or patients with known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Concurrent treatment with potent inhibitors of cytochrome P450 3A4, or patients planning to receive these treatments. For patients who were receiving treatment with such agents, a one-week washout period is required prior to registration.
* Peripheral neuropathy grade ≥ 2.
* Any of the following within the 6 months prior to registration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft surgery, clinically symptomatic and uncontrolled cardiovascular disease, or clinically significant cardiac arrhythmias (grade 3-4).
* History of inflammatory bowel disease or chronic diarrhea.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation or that may cause undue risk for the patient's safety.
* Known human immunodeficiency virus (HIV) infection requiring treatment or acquired immunodeficiency-syndrome (AIDS)-related illness.
* Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose (MTD) of XRP9881 when given in combination with capecitabine | study period

SECONDARY OUTCOMES:
Response in patients with measurable disease | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Paris, France